CLINICAL TRIAL: NCT01361750
Title: The Effects of Gastric Tube on the Quality of Life and Nutritional Status After Ivor-Lewis Esophagectomy: A Randomized Control Trial and Physiological Study
Brief Title: The Effects of Gastric Tube on the Quality of Life and Nutritional Status After Ivor-Lewis Esophagectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: higher occurrence of complication than expected for both groups
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Yang Yue, Thoracic Surgery II, Peking University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PKU-OES-001
Record Dates: First submitted 2011-05-24; First posted 2011-05-27 (Estimated); Last update posted 2020-03-31 (Actual); Status verified 2020-03

CONDITIONS: Oesophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Enteral Nutrition

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- gastirc tube group (Experimental): conduit will be perfomed by narrowed gastric tube
  Interventions: Procedure: gastric tube
- control group (No Intervention): conduit will be traditional subtotal stomach without any surgical modification

INTERVENTIONS:
Procedure: gastric tube — the stomach will be cut into a narrowed tube-shape conduit
  Arms: gastirc tube group

SUMMARY:
This study is to investigate the effects of narrowed gastric tube on postoperative nutritional status and the quality of life in esophageal cancer patients treated with Ivor-Lewis esopagectomy in a 12-month follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* esophageal cancer (squamous and adenocarcinoma subtypes)
* eligble for Ivor-Lowis esophagectomy
* expected survival time longer than 12 months

Exclusion Criteria:

* palliative resection(non-R0)
* anastomosis leak
* jejunum or colon transversum interponate

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-05; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
change of nutritional status and quality of life before and after operation | before operation (baseline), 1 month, 6 month and 12 month after operation

SECONDARY OUTCOMES:
change of serum markers and tissue inflammatory status before and after operation | before operation (baseline), 1 month, 6 month and 12 month after operation

CONTACTS AND LOCATIONS:
Overall Officials: Yue Yang, M.D., Principal Investigator — Peking University Health Science Center
Locations (1):
- Peking University School of Oncology, Beijing, Beijing Municipality, China